CLINICAL TRIAL: NCT00917241
Title: Prevention Relapse of Graves' Disease by Treatment With Intrathyroid Injection of Dexamethasone
Brief Title: Prevention Relapse of Graves' Disease by Intrathyroid Injection of Dexamethasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiao-Ming Mao (Other)
Responsible Party: Sponsor-Investigator, Xiao-Ming Mao, Professor, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NanjingMU
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2009-06

CONDITIONS: Graves' Disease
Keywords: Graves' disease; dexamethasone; relapse; methimazole
MeSH Terms: conditions — Graves Disease; Recurrence | interventions — Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMI+IID group (Experimental): MMI,methimazole；IID,intrathyroid injection of dexamethasone
  Interventions: Drug: MMI combined with IID
- MMI Group (Active Comparator): MMI,methimazole
  Interventions: Drug: MMI

INTERVENTIONS:
Drug: MMI combined with IID — MMI titration regimen for 18 months,initial dosage of MMI was 20 mg/d,which combined with IID for 3 months.Dexamethasone was injected into the two side of thyroid, the dose of dexamethasone was 5 mg by every side, twice a week. The treatment strategy was changed to once a week at the second month and twice a month at the third month, the dose of dexamethasone was the same as the first month.
  Other Names: methimazole,tapazole;dexamethasone,hexadecadrol
  Arms: MMI+IID group
Drug: MMI — MMI treatment with titration regimen for 18 months, initial dosage was 20 mg/d.
  Arms: MMI Group

SUMMARY:
Antithyroid drugs are widely used in treatment of Graves' disease (GD), but after therapy withdrawal, relapse rate is very high. The aim this trail is to evaluate the effects of intrathyroid injection of dexamethasone combined with antithyroid drugs on patients with newly diagnosed GD.

DETAILED DESCRIPTION:
The morbility of GD is nearly 0.5% and the underlying cause of 50 to 80% of cases of hyperthyroidism.Recently,anti-thyroid drugs are still the main therapy for Graves'hyperthyroidism in a lot of districts, but the relapse rate is very high (51~68%) after withdrawal of anti-thyroid treatment.In order to reduce the relapse rate, some studies tried to prescribe replacement thyroxine, either with the anti-thyroid drug treatment, or after this was completed, but there is no clear evidence in favour of giving thyroid hormone supplementation following the initial treatment of Graves' thyrotoxicosis with anti-thyroid medication. Therefore, the optimal medical therapy for Graves' hyperthyroidism remains a subject of debate.

It is well known that glucocorticoids have anti-inflammatory, immunomodulation and immunosuppression effects and they has long been used to treat GO, and is one of the most effective medicine ,it can decrease some cytokines and reduce inflammatory status ,and improve some thyroid specific antibody, like as thyrotropin receptor antibodies (TRAb), antithyroperoxidase antibodies (TPOAb) and antithyroglobulin antibodies (TGAb).These studies suggested that glucocorticoids might affect autoimmune process and have some benefit effects on GD. Moreover glucocorticoids have been used to treat GD in several early reports, in which serum free triiodothyronine (FT3) and thyroxine (FT4) or total T3(TT3) and TT4 levels decreased after 8 days or three weeks treatment with glucocorticoids . But in those studies, the number of selected patients is small, and the duration of the therapy is relatively short, so that might not confirm the effects of glucocorticoids on GD.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed of Graves' Disease

Exclusion Criteria:

* Pregnancy
* Allergy to ATD, Alanine aminotransferase (ALT) or asparate aminotransferase (AST) above 2 times of upper normal range
* Non-compliance because of psychiatric or other serious diseases, or unwillingness to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2004-06; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
relapse of hyperthyroidism | 4.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Mao, M.D., Principal Investigator — Affiliated Nanjing First Hospital, Nanjing Medical University

REFERENCES:
- [Derived] Mao XM, Li HQ, Li Q, Li DM, Xie XJ, Yin GP, Zhang P, Xu XH, Wu JD, Chen SW, Wang SK. Prevention of relapse of Graves' disease by treatment with an intrathyroid injection of dexamethasone. J Clin Endocrinol Metab. 2009 Dec;94(12):4984-91. doi: 10.1210/jc.2009-1252. Epub 2009 Oct 22. PMID 19850691